CLINICAL TRIAL: NCT07140601
Title: Environmental Pollutants and Neurological Disorders: Clinical and Mechanistic Study
Brief Title: Environmental Pollutants and Neurological Disorders
Acronym: CLEAN
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Chinese Research Academy of Environmental Sciences (Other); Nanjing University (Other); Nanjing Institute of Environmental Sciences (Unknown); Chinese Academy of Environmental Planning (Unknown); Peking Union Medical College (Other); National Human Brain Bank for Development and Function (Unknown)
Responsible Party: Principal Investigator, Xiaolin Chen, MD, Prof., Beijing Tiantan Hospital
Other Study IDs: KY2024-252-02; 2024ZD0539700 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-08-22; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebrovascular Disorders; Brain Tumours; Alzheimer Dementia
Keywords: Environmental Pollutants; Exposomics; Pathogenic Mechanisms; Neurological Disorders; Neurosurgical Patients
MeSH Terms: conditions — Cerebrovascular Disorders; Brain Neoplasms; Alzheimer Disease; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Environmental pollutants have emerged as a major global health concern, with growing evidence linking exposure to both traditional contaminants such as heavy metals (lead, mercury, cadmium, arsenic) and novel pollutants-including micro- and nanoplastics, per- and polyfluoroalkyl substances (PFAS), antibiotics, and endocrine-disrupting chemicals-to adverse neurological outcomes. These pollutants can cross or disrupt the blood-brain barrier, accumulate in neural tissue, and trigger oxidative stress, inflammation, epigenetic modifications, and metabolic reprogramming.

Brain tumours and cerebrovascular diseases represent two major categories of neurosurgical disorders with high morbidity and mortality. However, their interaction with environmental pollutant exposure remains poorly understood. Recent studies suggest that pollutant-induced molecular alterations, such as aberrant DNA methylation, lipid metabolism disruption, and neurovascular endothelial dysfunction, may contribute to tumour initiation, malignant progression, aneurysm formation, and stroke occurrence.

Given the increasing human exposure to these pollutants and the lack of large-scale clinical data, it is urgent to establish a systematic investigation in neurosurgical patients. This study aims to profile pollutant exposure (heavy metals, PFAS, microplastics, and other novel contaminants) using multi-biospecimen analysis (blood, urine, hair, tumour and peri-tumour tissues), and to explore their mechanistic links to the pathogenesis of brain tumours and cerebrovascular diseases. The findings are expected to provide new evidence for understanding environment-brain interactions and to identify potential biomarkers for disease risk stratification and prevention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Able to give informed consent to participate in the research.

Exclusion Criteria:

* Refusal to participate.
* Pregnant or breastfeeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with brain tumours or cerebrovascular diseases who need surgical resection.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Until death or study completion (24 months)
  OS is defined as the time from the sample collection date to death due to any cause. All other participants will be censored at the last date known to be alive.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Until progression or death or study completion (24 months)
  PFS is defined as the duration of time from sample collection date to time of progression or death, whichever occurs first.
modified Rankin Scale (mRS) | 90 days after sample collection
  Patients' mRS scores at 90 days after sample collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided